CLINICAL TRIAL: NCT00807729
Title: Prospective Randomized Trial of Laparoscopic Cholecystectomy Plus Laparoscopic Common Bile Duct Exploration (LC + LCBDE) Versus Endoscopic Retrograde Cholangiopancreatography Sphincterotomy Plus Laparoscopic Cholecystectomy (ERCP/S + LC) for Common Bile Duct Stone Disease
Brief Title: Randomized Trial of ERCP Then Laparoscopic Cholecystectomy vs. Laparoscopic Cholecystectomy Plus Laparoscopic Common Bile Duct Exploration in Patients With Likely Choledocholithiasis
Acronym: ERCP/CBDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Stanley J. Rogers, MD - Associate Professor of Surgery, UCSF, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H9437-10261-12; K08DK002607 (NIH)
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Choleclithiasis; Common Bile Duct Stones
Keywords: Laparoscopy; Endoscopic retrograde cholangiopancreatography; Sphincterotomy; Common bile duct stones; Laparoscoopic common bile duct exploration; Cost efficiency; Examination of efficacy, safety, cost of intervention for patients with choleclithiasis and likely common bile duct stones
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde; Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERCP (Active Comparator): All ERCP's were performed by one of the authors (JPC), a fulltime faculty member and gastroenterology fellowship instructor in the presence and concurrence of the principal author/ surgeon (SJR). Patients randomized to ERCP/S + LC were scheduled to undergo the endoscopic procedure using fluoroscopy (OEC Diasonics 9400) in the endoscopy suite under moderate sedation (principally intravenous midazolam and meperidine) prior to the intended laparoscopy. Duodenal atony during ERCP was routinely achieved using intravenout glucagon. The laparoscopic cholecystectomy was subsequently performed as soon as technically feasible (i.e. following abdominal gas decompression) following the ERCP
  Interventions: Procedure: ERCP
- Lap CBDE (Active Comparator): LC + LCBDE was performed in a routine fashion by one fulltime faculty member (SJR) with fellowship training in laparoscopy. Cholangiograms were obtained fluoroscopically using the same make and model fluoroscope (OEC Diasonics 9400) as used in ERCP by antegrade contrast flushing through the cystic duct. All fluoroscopy was performed by the principal author (SJR) in the presence of and concurrence with the ERCP endoscopist (JPC). When stones were detected or suspected by cholangiography, transcystic exploration was undertaken by balloon or basket with associated balloon dilation of the sphincter of Oddi A completion cholangiogram was obtained to confirm that all stones were removed. Once the LCBDE was completed, the cystic duct was ligated and the gallbladder removed.
  Interventions: Procedure: LapCBDE

INTERVENTIONS:
Procedure: ERCP — Endoscopic Retrograde Cholangiopancreatography Patients randomized to ERCP/S + LC were scheduled to undergo the endoscopic procedure using fluoroscopy (OEC Diasonics 9400) in the endoscopy suite under moderate sedation (principally intravenous midazolam and meperidine) prior to the intended laparoscopy. Duodenal atony during ERCP was routinely achieved using intravenout glucagon. If choledocholithiasis was detected or suspected at the time of ERCP, a sphincterotomy was undertaken so that gallstones could be extracted using a balloon catheter or retrieval basket. Small bowel gas was aspirated endoscopically as much as possible at the conclusion of the ERCP. The laparoscopic cholecystectomy was subsequently performed as soon as technically feasible (i.e. following abdominal gas decompression) following the ERCP
  Other Names: ERCP/ laparoscopic cholecystectomy
  Arms: ERCP
Procedure: LapCBDE — LC + LCBDE was performed in a routine fashion by one fulltime faculty member (SJR) with fellowship training in laparoscopy. Cholangiograms were obtained fluoroscopically using the same make and model fluoroscope (OEC Diasonics 9400) as used in ERCP by antegrade contrast flushing through the cystic duct. All fluoroscopy was performed by the principal author (SJR) in the presence of and concurrence with the ERCP endoscopist (JPC). When stones were detected or suspected by cholangiography, transcystic exploration was undertaken by balloon or basket with associated balloon dilation of the sphincter of Oddi A completion cholangiogram was obtained to confirm that all stones were removed. Once the LCBDE was completed, the cystic duct was ligated and the gallbladder removed.
  Other Names: Laparoscopic common bile duct exploration
  Arms: Lap CBDE

SUMMARY:
Objective: We compared outcome parameters for good-risk patients with classic signs, symptoms, laboratory and abdominal imaging features of cholecystolithiasis and choledocholithiasis randomized to either LC + LCBDE or ERCP/S + LC.

Design: Our study was a prospective trial conducted following written informed consent with randomization by the serially-numbered opaque envelope technique.

Setting: Our institution is an academic teaching hospital and the central receiving and trauma center for the City and County of San Francisco.

Patients: We randomized 122 patients (American Society of Anesthesiologists Grade I or II) meeting entry criteria. Ten of these patients, excluded from outcome analysis, were protocol violators having signed out of the hospital against medical advice before one of both procedures were completed.

Interventions: Treatment was pre-operative endoscopic retrograde cholangiopancreatography sphincterotomy (ERCP/S) followed by laparoscopic cholecystectomy (LC), or laparoscopic cholecystectomy plus laparoscopic common bile duct exploration (LC + LCBDE).

Main Outcome Measures: The primary outcome measure was efficacy of stone clearance from the common bile duct. Secondary endpoints were length of hospital stay, cost of index hospitalization, professional fees, hospital charges, morbidity and mortality, and patient acceptance and quality of life scores.

DETAILED DESCRIPTION:
Objective: We compared outcome parameters for good-risk patients with classic signs, symptoms, laboratory and abdominal imaging features of cholecystolithiasis and choledocholithiasis randomized to either LC + LCBDE or ERCP/S + LC.

Design: Our study was a prospective trial conducted following written informed consent with randomization by the serially-numbered opaque envelope technique.

Setting: Our institution is an academic teaching hospital and the central receiving and trauma center for the City and County of San Francisco.

Patients: We randomized 122 patients (American Society of Anesthesiologists Grade I or II) meeting entry criteria. Ten of these patients, excluded from outcome analysis, were protocol violators having signed out of the hospital against medical advice before one of both procedures were completed.

Interventions: Treatment was pre-operative endoscopic retrograde cholangiopancreatography sphincterotomy (ERCP/S) followed by laparoscopic cholecystectomy (LC), or laparoscopic cholecystectomy plus laparoscopic common bile duct exploration (LC + LCBDE).

Main Outcome Measures: The primary outcome measure was efficacy of stone clearance from the common bile duct. Secondary endpoints were length of hospital stay, cost of index hospitalization, professional fees, hospital charges, morbidity and mortality, and patient acceptance and quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Classic biliary-type pain
* Ultrasonographic demonstration of cholecystolithiasis
* Platelet count > 100,000 per mm³ and prothrombin time < 3 seconds of control
* American Society of Anesthesiology (ASA) risk grade I or II:

  1. Common bile duct diameter greater than 6 mm by ultrasound or computed tomography (CT) scan
  2. Intrahepatic duct dilation as determined by ultrasound or CT scan Serum bilirubin greater than 2mg/dl, alkaline phosphatase and/or lipase more than 1.5 times upper limit of normal within 48 hours of intended first pro

Exclusion Criteria:

* History of bleeding disorders, platelet count <100,000 per mm³ and/or prothrombin time >3 seconds over control
* Uremia as evidenced by a creatinine > 3 mg/dl and/or blood urea nitrogen > 50 mg/dl
* Ultrasonography or CT evidence of cirrhosis, intrahepatic gallbladder, liver mass or abscess, or periampullary neoplasm
* Insulin-dependent diabetes mellitus
* Multiple prior laparotomies
* Morbid obesity
* Clinical, radiologic and/or biochemical evidence of cirrhosis or portal vein thrombosis
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 1997-01; Primary Completion 2003-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the efficacy of common bile duct stone clearance. | Hospital admmission

SECONDARY OUTCOMES:
Secondary endpoints were length of hospital stay, total cost of index hospitalization, professional fee charges, hospital charges, morbidity and mortality, and patient acceptance and quality of life scores. | Hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Rogers SJ, Cello JP, Horn JK, Siperstein AE, Schecter WP, Campbell AR, Mackersie RC, Rodas A, Kreuwel HT, Harris HW. Prospective randomized trial of LC+LCBDE vs ERCP/S+LC for common bile duct stone disease. Arch Surg. 2010 Jan;145(1):28-33. doi: 10.1001/archsurg.2009.226. PMID 20083751